CLINICAL TRIAL: NCT04003259
Title: Comprehensive Lifestyle Management Programme in the Treatment of Obesity: the Get-a-Grip (GAG) Study
Brief Title: Get-a-Grip Lifestyle Management Programme
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tampere University (Other)
Collaborators: Tampere University Hospital (Other); Sitra, the Finnish Innovation Fund (Other)
Responsible Party: Principal Investigator, Ilkka Pörsti, MD, Clinical Professor, Tampere University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R12099
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Overweight and Obesity; Hypertension; Dyslipidemias; Diabetes
Keywords: Diet; Exercise; Lifestyle; Weight control
MeSH Terms: conditions — Overweight; Obesity; Hypertension; Dyslipidemias; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Overweight and obese subjects (Experimental): 1-year lifestyle programme
  Interventions: Behavioral: Lifestyle management programme

INTERVENTIONS:
Behavioral: Lifestyle management programme — The programme consisted of 1) the initiation phase (1-3 months), 2) the establishment phase (3-6 months), and 3) the maintenance phase (7-12 months). Guidance was given altogether on 25 separate occasions with special emphasis on the motivation and education. The goal for weight loss was 5-10 %. The programme included four visits by medical doctor, an educational lecture by medical doctor and personal trainer, five sessions by registered dietician, two cooking classes by professional chef, two group discussions, and exercise as follows: personalized exercise program tailored by personal trainer, one-year gym access with four guided group sessions, and two guided group Nordic walking sessions, and three individual exercise sessions by personal trainer.

SUMMARY:
The primary aim of this study was to examine weight reduction in primary care in obese or overweight subjects with a comorbidity that would benefit from weight loss during 1-year comprehensive lifestyle management programme including medical examinations, personalized dietary and exercise advice, guidance on shopping behaviour and food preparation, and group discussions.

DETAILED DESCRIPTION:
Obesity is associated with altered glucose and lipid metabolism, and elevated blood pressure (BP) increasing the risk of cardiovascular morbidity and mortality. Obesity-induced complications are increasingly encountered in the health care system and especially in primary care. Thus, there is a growing need for individually tailored weight management programs aiming to permanent lifestyle and dietary changes for the prevention and treatment of obesity-related health hazards.

The study investigated weight reduction during 1-year comprehensive lifestyle programme in 134 obese or overweight subjects (BMI>30, or BMI>25 with a comorbidity including diabetes, hypertension, arthrosis, asthma, chronic obstructive lung disease, sleep apnoea). The participants were recruited from the local diabetes centre and health care providers. The programme aimed at 5-10 % weight reduction utilizing exercise program supervised by personal trainer, advice on diet and on-location shopping behavior by a registered dietician, hands-on cooking classes by a professional chef, examinations by a medical doctor, and group discussions. The efficacy of the program was followed by measuring change in weight, BMI, waist circumference, fat and muscle percentage, visceral fat, and systolic and diastolic BP.

The study protocol has been approved by the ethics committee of the Pirkanmaa Hospital District (R12099).

ELIGIBILITY:
Inclusion Criteria:

* BMI >30
* BMI>25 with a co-morbidity that would benefit from weight loss (diabetes, hypertension, arthrosis, asthma, chronic obstructive lung disease, sleep apnoea)

Exclusion Criteria:

* physical condition that prevented exercise
* abuse of alcohol or drugs
* medical history suggesting poor adherence
* severe concurrent disease
* moderate to severe dementia

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2009-01-01 (Actual); Primary Completion 2013-12-31 (Actual); Study Completion 2013-12-31 (Actual)

PRIMARY OUTCOMES:
Change in weight (kg) | baseline, and months 2-3, 5-6, and 11-12
  Weight was measured at baseline (month 0), and after 2-3, 5-6, and 11-12 months.
Change in body mass index (BMI) (kg/m^2) | baseline, and months 2-3, 5-6, and 11-12
  BMI was measured at baseline (month 0), and after 2-3, 5-6, and 11-12 months.
Change in waist circumference (cm) | baseline, and months 2-3, 5-6, and 11-12
  Waist circumference was measured at baseline (month 0), and after 2-3, 5-6, and 11-12 months.
Change in muscle mass and body fat (percentage points) | baseline, and months 2-3, 5-6, and 11-12
  Muscle and fat percentage were measured at baseline (month 0), and after 2-3, 5-6, and 11-12 months.
Change in systolic and diastolic blood pressure (mmHg) | baseline, and months 2-3, 5-6, and 11-12
  Blood pressure was measured at baseline (month 0), and after 2-3, 5-6, and 11-12 months.

SECONDARY OUTCOMES:
Fitness index | All participants were invited to a two-kilometer walk-test at baseline (month 0) and month 11-12
  Fitness index was constructed from a two-kilometer walk test with heart rate monitoring and took into consideration age, gender, height, weight, walking time, and heart rate.

CONTACTS AND LOCATIONS:
Overall Officials: Ilkka Pörsti, MD, PhD, Principal Investigator — Tampere University
Locations (1):
- Tampere University Hospital, Tampere, Southern Finland, Finland

IPD SHARING:
Plan to Share IPD: No
Analyses and generated datasets during the current study are not available publicly as the informed consent obtained does not allow publication of individual patient data. However, raw data is available from the principal investigator (email ilkka.porsti@tuni.fi) on reasonable request.

REFERENCES:
- [Derived] Taurio J, Jarvinen J, Hautaniemi EJ, Eraranta A, Viitala J, Nordhausen K, Kaukinen K, Mustonen J, Porsti IH. Team-based "Get-a-Grip" lifestyle management programme in the treatment of obesity. Prev Med Rep. 2020 May 13;19:101119. doi: 10.1016/j.pmedr.2020.101119. eCollection 2020 Sep. PMID 32461881